CLINICAL TRIAL: NCT04083976
Title: A Phase 2 Study of Erdafitinib in Subjects With Advanced Solid Tumors and FGFR Gene Alterations
Brief Title: A Study of Erdafitinib in Participants With Advanced Solid Tumors and Fibroblast Growth Factor Receptor (FGFR) Gene Alterations
Acronym: RAGNAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108661; 42756493CAN2002 (Other: Janssen Research & Development, LLC); 2019-002113-19 (EudraCT Number); 2023-510301-18-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erdafitinib (Experimental): Participants with fibroblast growth factor receptor (FGFR) mutations and FGFR gene fusions will receive a dose of erdafitinib oral tablets until disease progression, intolerable toxicity, withdrawal of consent, decision by the investigator to discontinue treatment, or end of data collection timepoint if there is clinical benefit in the opinion of the investigator, has been achieved.
  Interventions: Drug: Erdafitinib

INTERVENTIONS:
Drug: Erdafitinib — Participants will receive erdafitinib oral tablets.
  Other Names: JNJ-42756493

SUMMARY:
The purpose of this study is to evaluate the efficacy of erdafitinib in terms of overall response rate (ORR) in adult and pediatric participants with advanced solid tumors with fibroblast growth factor receptor (FGFR) alterations (mutations or gene fusions). It will also evaluate ORR in pediatric participants with advanced solid tumors and FGFR alterations.

DETAILED DESCRIPTION:
Erdafitinib is a selective and potent pan FGFR 1-4 inhibitor with demonstrated clinical activity in participants with metastatic urothelial cancer and cholangiocarcinoma identified to have alterations in the FGFR pathway. This study targets the underlying altered biology of FGFR-driven tumors irrespective of solid tumor histology subtype. The study consists of screening phase, treatment phase and the post treatment follow-up phase (from the end of treatment visit until the participant has died, withdraws consent, is lost to follow-up, or the end of study, whichever comes first). End of study is considered as the time when the last participant receives the last dose of study drug on the study and either all pediatric participants are off study or until the most recently enrolled pediatric participant still participating in the study has 6 months of follow-up, whichever occurs first. Currently this study is recruiting pediatric participants only.

ELIGIBILITY:
Inclusion Criteria:

* Histologic demonstration of an unresectable, locally advanced, or metastatic solid tumor malignancy with an fibroblast growth factor receptor (FGFR) mutation or FGFR gene fusion
* Measurable disease
* Participant must have received at least one prior line of systemic therapy in the advanced, unresectable, or metastatic setting; or is a child or adolescent participant with a newly-diagnosed solid tumor and no acceptable standard therapies
* Documented progression of disease, defined as any progression that requires a change in treatment, prior to full study screening

Exclusion Criteria:

* Has had prior chemotherapy, targeted therapy, or treatment with an investigational anticancer agent within 15 days or less than or equal to (<=) 5 half-lives of the agent (whichever is longer) and up to a maximum of 30 days before the first dose of erdafitinib
* The presence of FGFR gatekeeper and resistance mutations
* Histologic demonstration of urothelial carcinoma
* Hematologic malignancy (i.e., myeloid and lymphoid neoplasms
* For non-small cell lung cancer participants only: pathogenic somatic mutations or gene fusions in the following genes: EGFR, ALK, ROS1, NTRK, BRAF V600E and KRAS
* Active malignancies other than for disease requiring therapy

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (171):
- United States (27):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Memorial Cancer Institute, Hollywood, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Hawaii Cancer Care, ‘Aiea, Hawaii
  - Maine Medical Center, Scarborough, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - MD Anderson, Houston, Texas
  - Oncology Consultants Texas, Houston, Texas
  - Texas Oncology Odessa-West Texas Cancer Center, Odessa, Texas
  - Texas Oncology San Antonio Northeast, San Antonio, Texas
  - NorthWest Medical Specialties, PLLC, Tacoma, Washington
  - Aurora Research Institute, Wauwatosa, Wisconsin
- Argentina (12):
  - Instituto de Investigaciones Metabólicas, Buenos Aires
  - Hospital Aleman, Buenos Aires
  - Centro Oncológico Korben, Buenos Aires
  - Instituto Fleni, Buenos Aires
  - CEMIC Saavedra, Buenos Aires
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Hospital Italiano de La Plata, La Plata Lpl Lpl
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Hospital Privado de Comunidad, Mar del Plata
  - Hospital Universitario Austral, Pilar
  - Sanatorio Britanico de Rosario, Rosario
  - ARS Médica, San Salvador de Jujuy
- Australia (6):
  - Flinders Centre for Innovation in Cancer, Adelaide
  - Chris O'Brien Lifehouse, Camperdown
  - St Vincent s Hospital Sydney, Darlinghurst
  - St Vincents Hospital Melbourne, Fitzroy
  - Fiona Stanley Hospital, Murdoch
  - Intergrated Clinical Oncology Network Pty Ltd (ICON), South Brisbane
- Belgium (11):
  - AZ Klina, Brasschaat
  - UCL Hopital Saint-Luc, Brussels
  - Grand Hopital de Charleroi, site Notre Dame, Charleroi
  - CHU UCL Namur - Site Dinant, Dinant
  - UZA, Edegem
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - Jolimont, Haine-Saint-Paul
  - CHU UCL Namur - Site Sainte Elisabeth, Namur
  - Cliniques St Pierre, Ottignies
  - CHU UCL Namur - Site Godinne, Yvoir
- Brazil (16):
  - Fundacao Pio XII, Barretos
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Associacao de Combate ao Cancer em Goias - Hospital de Cancer Araujo Jorge, Goiânia
  - Associacao Hospital de Caridade Ijui, Ijuí
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
  - GRAACC, São Paulo
- China (18):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - Jilin cancer hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - West China Hospital,Sichuan University, Chengdu
  - Chongqing Southwest Hospital, Chongqing
  - Third Military Medical University Daping Hospital Cancer Center, Chongqing
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Eastern Theater General Hospital, Qinhuai District Medical Area, Nanjing
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Cancer Hospital, FuDan University, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Huashan Hospital Fudan University, Shanghai
- France (11):
  - Hopital Saint André, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital de la Timone, Marseille
  - Institut Curie, Paris
  - CHU De Poitiers, Poitiers
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (11):
  - Charité, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Medizinische Fakultaet Carl Gustav Carus Technische Universitaet Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Asklepios Klinik Altona, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Klinikum rechts der Isar der TU Munchen, München
  - Universitatsklinikum Tubingen, Tübingen
- Italy (9):
  - Istituto Ortopedico Rizzoli, Bologna
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - ASST di Monza, Monza
  - Azienda Ospedaliera Univ.- Università Degli studi della Campania - Luigi Vanvitelli, Napoli
  - Fondazione G Pascale Istituto Nazionale Tumori IRCCS, Napoli
  - Ospedale S. Maria Della Misericordia, Perugia
  - Ospedale Santa Chiara AO Universitaria Pisana, Pisa
  - Azienda Ospedaliera S. Maria Terni, Terni
  - Ospedale Borgo Roma, Verona
- Japan (5):
  - National Cancer Center Hospital, Chūōku
  - Hiroshima University Hospital, Hiroshima
  - National Cancer Center Hospital East, Kashiwa
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Fujita Health University Hospital, Toyoake
- Poland (8):
  - Centrum Onkologii im Prof F Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Instytut Matki i Dziecka, Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- South Korea (5):
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (13):
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Sant Joan de Deu, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, L'Hospitalet de Llobregat
  - Hosp. Infantil Univ. Nino Jesus, Madrid
  - Clinica Univ. de Navarra, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- Taiwan (12):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - E-Da Cancer Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center Yong Kang, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center Liu Ying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan
- United Kingdom (7):
  - Bristol Royal Hospital for Children, Bristol
  - Bristol Haematology and Oncology Centre, Bristol
  - The Christie Nhs Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle upon Tyne
  - Derriford Hospital, Plymouth
  - The Royal Marsden NHS Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Pant S, Schuler M, Iyer G, Witt O, Doi T, Qin S, Tabernero J, Reardon DA, Massard C, Minchom A, Lugowska I, Carranza O, Arnold D, Gutierrez M, Winter H, Stuyckens K, Crow L, Najmi S, Hammond C, Thomas S, Santiago-Walker A, Triantos S, Sweiti H, Loriot Y; RAGNAR Investigators. Erdafitinib in patients with advanced solid tumours with FGFR alterations (RAGNAR): an international, single-arm, phase 2 study. Lancet Oncol. 2023 Aug;24(8):925-935. doi: 10.1016/S1470-2045(23)00275-9. PMID 37541273

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As pre-specified in the protocol, adolescent participants enrolled in the Broad Panel Cohort who met the pediatric cohort definition were planned to be analyzed as part of the Broad Panel Cohort and the Pediatric Cohort. 2 adolescent participants from the broad panel cohort were included in the pediatric cohort. Hence, these 2 participants are counted as enrolled twice (once in Broad Panel Cohort and once in Pediatric Cohort).
Groups:
- Broad Panel Cohort: Adolescent and adult participants with target fibroblast growth factor receptor (FGFR) mutations or any FGFR gene fusions, were enrolled in this cohort. Adolescent participants aged greater than or equal to (>=)12 to less than (<)15 years received erdafitinib 5 milligrams (mg) once daily orally, with possible up-titration to 6 mg or further to 8 mg based on Cycle 1 Day 14 and Cycle 2 Day 7 (each cycle of 21 days) serum phosphate levels. Adolescent participants aged >=15 to <18 years and adults participants aged 18 years and older received erdafitinib 8 mg once daily orally, with possible up-titration to 9 mg or maintenance at 8 mg daily based on Cycle 1 Day 14 serum phosphate levels.
- Cholangiocarcinoma (CCA) Expansion Cohort: Adolescent and adult participants with target FGFR mutations or any FGFR gene fusion once the broad panel cohort has reached the cap of approximately 30 participants for cholangiocarcinoma, were enrolled in this cohort. Adolescent participants aged >=12 to <15 years received erdafitinib 5 mg once daily orally, with possible up-titration to 6 mg or further to 8 mg based on Cycle 1 Day 14 and Cycle 2 Day 7 (each cycle of 21 days) serum phosphate levels. Adolescent participants aged >=15 to <18 years and adults participants aged 18 years and older received erdafitinib 8 mg once daily orally, with possible up-titration to 9 mg or maintenance at 8 mg daily based on Cycle 1 Day 14 serum phosphate levels.
- Exploratory Cohort: Adolescent and adult participants with any other FGFR mutations that are not captured in the broad panel cohort, were enrolled in this cohort. Adolescent participants aged >=12 to <15 years received erdafitinib 5 mg once daily orally, with possible up-titration to 6 mg or further to 8 mg based on Cycle 1 Day 14 and Cycle 2 Day 7 (each cycle of 21 days) serum phosphate levels. Adolescent participants aged >=15 to <18 years and adults participants aged 18 years and older received erdafitinib 8 mg once daily orally, with possible up-titration to 9 mg or maintenance at 8 mg daily based on Cycle 1 Day 14 serum phosphate levels.
- Pediatric Cohort: Children and adolescent (from Broad Panel cohort) participants with locally advanced or metastatic solid tumors harboring FGFR alterations, any gene fusions or FGFR internal tandem duplication who had either progressed on prior therapies and who had no acceptable standard therapies, or who had a newly diagnosed solid tumor and who had no acceptable standard therapies, were enrolled in this cohort. Children aged >=6 to <12 years received erdafitinib 3 mg once daily orally with possible up-titration to 4 mg or further to 5 mg based on Cycle 1 Day 14 and Cycle 2 Day 7 (each cycle of 21 days) serum phosphate levels. Adolescent participants aged >=12 to <15 years received erdafitinib 5 mg once daily orally, with possible up-titration to 6 mg or further to 8 mg based on Cycle 1 Day 14 and Cycle 2 Day 7 serum phosphate levels, Adolescent participants aged >=15 to <18 years received erdafitinib 8 mg once daily orally, with possible up-titration to 9 mg or maintenance at 8 mg daily based on Cycle 1 Day 14 serum phosphate levels.
Period: Overall Study
Arm/Group | Broad Panel Cohort | Cholangiocarcinoma (CCA) Expansion Cohort | Exploratory Cohort | Pediatric Cohort
Started | 217 | 35 | 53 | 11
Adolescent Participants From Broad Panel Cohort | 0 | 0 | 0 | 2
Core Panel Cohort (Sub-group of Broad Panel Cohort) | 109 | 0 | 0 | 0
Completed | 183 | 34 | 43 | 3
Not Completed | 34 | 1 | 10 | 8
Not completed — Lost to Follow-up | 3 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 16 | 1 | 9 | 0
Not completed — Sponsor Decision | 14 | 0 | 0 | 7
Not completed — Other | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 2 adolescent participants from the broad panel cohort who were included in the pediatric cohort were analyzed in both broad panel cohort and pediatric cohort as planned.
Groups:
- Pediatric Cohort: Children and adolescent (from Broad Panel cohort) participants with locally advanced or metastatic solid tumors harboring FGFR alterations, any gene fusions or FGFR internal tandem duplication who had either progressed on prior therapies and who had no acceptable standard therapies, or who had a newly diagnosed solid tumor and who had no acceptable standard therapies, were enrolled in this cohort. Children aged >=6 to <12 years received erdafitinib 3 mg once daily orally, with possible up-titration to 4 mg or further to 5 mg based on Cycle 1 Day 14 and Cycle 2 Day 7 (each cycle of 21 days) serum phosphate levels. Adolescent participants aged >=12 to <15 years received erdafitinib 5 mg once daily orally, with possible up-titration to 6 mg or further to 8 mg based on Cycle 1 Day 14 and Cycle 2 Day 7 serum phosphate levels, Adolescent participants aged >=15 to <18 years received erdafitinib 8 mg once daily orally, with possible up-titration to 9 mg or maintenance at 8 mg daily based on Cycle 1 Day 14 serum phosphate levels.
- Total: Total of all reporting groups
Arm/Group | Broad Panel Cohort | Cholangiocarcinoma (CCA) Expansion Cohort | Exploratory Cohort | Pediatric Cohort | Total
Number analyzed (Participants) | 217 | 35 | 53 | 11 | 316
Age, Customized [Count of Participants; unit: Participants]
  6 years to <12 years | 0 | 0 | 0 | 4 | 4
  12 years to <18 years | 2 | 0 | 0 | 7 | 9
  18 years to <65 years | 162 | 25 | 31 | 0 | 218
  65 years and over | 53 | 10 | 22 | 0 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 23 | 32 | 7 | 159
  Male | 120 | 12 | 21 | 4 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 1 | 0 | 5 | 15
  Not Hispanic or Latino | 173 | 27 | 52 | 4 | 256
  Unknown or Not Reported | 35 | 7 | 1 | 2 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 57 | 11 | 24 | 2 | 94
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 6 | 0 | 4 | 2 | 12
  White | 112 | 18 | 25 | 5 | 160
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 38 | 6 | 0 | 2 | 46
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 2 | 0 | 0 | 4 | 6
  AUSTRALIA | 12 | 2 | 4 | 0 | 18
  BELGIUM | 10 | 5 | 7 | 0 | 22
  BRAZIL | 8 | 1 | 0 | 1 | 10
  CHINA | 12 | 3 | 0 | 0 | 15
  FRANCE | 26 | 5 | 0 | 1 | 32
  GERMANY | 22 | 4 | 4 | 0 | 30
  ITALY | 3 | 0 | 0 | 0 | 3
  JAPAN | 23 | 3 | 2 | 2 | 30
  POLAND | 3 | 0 | 3 | 0 | 6
  SOUTH KOREA | 6 | 1 | 7 | 0 | 14
  SPAIN | 16 | 3 | 6 | 1 | 26
  TAIWAN | 12 | 4 | 15 | 0 | 31
  UNITED KINGDOM | 14 | 1 | 4 | 0 | 19
  UNITED STATES | 48 | 3 | 1 | 2 | 54
AgeContinuous [Mean (Standard Deviation); unit: years] | 55.6 (13.51) | 57 (9.94) | 60 (11.74) | 12.4 (2.98) | 55 (15.07)

OUTCOME MEASURES:

1. Primary Outcome: Broad Panel and Pediatric Cohorts: Objective Response Rate (ORR) Based on Response Assessment in Neuro-Oncology (RANO) as Assessed by Independent Review Committee (IRC)
Description: ORR is defined as the percentage of participants who achieved a complete response (CR), or partial response (PR) based on Response Assessment in Neuro-Oncology (RANO) criteria. According to RANO criteria whereby overall RANO response is based on both radiographic response (CR: disappearance of all target lesions; PR: sum of products of diameters [SPD] decreased by >=50 percent [%] from baseline value) and clinical performance status with steroid dose information.
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 4 years
Population: The treated population consisted of all participants in broad panel and pediatric cohorts who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Broad Panel Cohort | Pediatric Cohort
Number analyzed (Participants) | 217 | 3
Percentage of participants | 29.5 [23.5 to 36.0] | 66.7 [9.4 to 99.2]

2. Primary Outcome: Core Panel Cohort: Objective Response Rate (ORR) Based on Response Assessment in Neuro-Oncology (RANO) as Assessed by Independent Review Committee (IRC)
Description: ORR is defined as the percentage of participants who achieved a CR, or PR based on RANO criteria. According to RANO criteria whereby overall RANO response is based on both radiographic response (CR: disappearance of all target lesions; PR: sum of products of diameters [SPD] decreased by >=50 percent [%] from baseline value) and clinical performance status with steroid dose information. The core panel cohort is a subgroup of the broad panel cohort with a select panel of pre-specified FGFR markers: FGFR3 mutations (S249C;Y373C; R248C; G370C); FGFR2 mutations (C382R); FGFR3 fusions (FGFR3-TACC3); FGFR2 fusions (FGFR2-BICC1; FGFR2-TACC2).
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 4 years
Population: The treated population (core panel) consisted of a subgroup of participants in the broad panel cohort (fibroblast growth factor receptor [FGFR+]) with a select panel of pre-specified FGFR markers who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Core Panel Cohort: Core panel cohort is a sub-group of broad panel cohort. Adolescent and adult participants with target FGFR mutations or any FGFR gene fusions, were enrolled in this cohort. Adolescent participants aged >=12 to <15 years received erdafitinib 5 mg once daily orally, with possible up-titration to 6 mg or further to 8 mg based on Cycle 1 Day 14 and Cycle 2 Day 7 serum phosphate levels. Adolescent participants aged >=15 to <18 years and adults participants aged 18 years and older received erdafitinib 8 mg once daily orally, with possible up-titration to 9 mg or maintenance at 8 mg daily based on Cycle 1 Day 14 serum phosphate levels.
Arm/Group | Core Panel Cohort
Number analyzed (Participants) | 109
Percentage of participants | 26.6 [18.6 to 35.9]

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Investigators Assessment
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

4. Secondary Outcome: Duration of Responses (DOR)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

5. Secondary Outcome: Disease Control Rate (DCR)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Clinical Benefit Rate (CBR)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

7. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

8. Secondary Outcome: Overall Survival (OS)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) by Severity
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

11. Secondary Outcome: Pediatric Cohort: Plasma Concentration of Erdafitinib
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

12. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) for Participants >=18 Years
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

13. Secondary Outcome: Change From Baseline in Pediatric Functional Assessment Of Cancer Therapy-Brain (Peds FACT-Br)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

14. Secondary Outcome: Change From Baseline in Patient Global Impression of Symptom Severity (PGIS)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

15. Secondary Outcome: Change From Baseline in Patient Global Impression of Change (PGIC)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

16. Secondary Outcome: Change From Baseline in European Quality of Life -5 Dimensions-5 Levels (EQ-5D-5L)
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 5 years 4 months
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: Baseline (Cycle 1 Day 1 [each cycle of 21 days]) up to 4 years
Description: The treated population consisted of all participants (FGFR+) who received at least 1 dose of study drug. 2 adolescent participants from the broad panel cohort who were included in the pediatric cohort were analyzed in both broad panel cohort and pediatric cohort as planned.
Arm/Group | Broad Panel Cohort | Cholangiocarcinoma (CCA) Expansion Cohort | Exploratory Cohort | Pediatric Cohort
All-Cause Mortality (participants affected / at risk) | 8/217 | 1/35 | 1/53 | 1/11
Serious Adverse Events (participants affected / at risk) | 86/217 | 15/35 | 26/53 | 8/11
Other Adverse Events (participants affected / at risk) | 215/217 | 35/35 | 53/53 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Broad Panel Cohort (N=217) | Cholangiocarcinoma (CCA) Expansion Cohort (N=35) | Exploratory Cohort (N=53) | Pediatric Cohort (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral Valve Stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 0 | 0
Chorioretinopathy (Eye disorders) | 0 | 1 | 0 | 0
Corneal Epithelium Defect (Eye disorders) | 0 | 0 | 1 | 0
Corneal Oedema (Eye disorders) | 0 | 0 | 1 | 0
Detachment of Retinal Pigment Epithelium (Eye disorders) | 0 | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 1 | 0
Keratitis (Eye disorders) | 0 | 2 | 0 | 0
Retinal Oedema (Eye disorders) | 1 | 0 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 8 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anal Erosion (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric Stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Malignant Gastrointestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Obstruction Gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 0 | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Asthenia (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0
Gait Disturbance (General disorders) | 1 | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 5 | 0 | 2 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 0 | 0
Performance Status Decreased (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 6 | 0 | 1 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary Dilatation (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 3 | 2 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatobiliary Disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic Shock (Immune system disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Biliary Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 2 | 0 | 0 | 0
Escherichia Infection (Infections and infestations) | 1 | 0 | 0 | 0
Liver Abscess (Infections and infestations) | 1 | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 0 | 1 | 0
Pseudomonas Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 1
Tooth Infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
General Physical Condition Abnormal (Investigations) | 1 | 0 | 0 | 0
Liver Function Test Increased (Investigations) | 1 | 0 | 0 | 0
Pulse Absent (Investigations) | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Brain Stem Infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Intraventricular Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Partial Seizures (Nervous system disorders) | 1 | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 2 | 0 | 0 | 0
Status Epilepticus (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0
Vasogenic Cerebral Oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 4 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Broad Panel Cohort (N=217) | Cholangiocarcinoma (CCA) Expansion Cohort (N=35) | Exploratory Cohort (N=53) | Pediatric Cohort (N=11)
Anaemia (Blood and lymphatic system disorders) | 57 | 13 | 9 | 3
Leukopenia (Blood and lymphatic system disorders) | 12 | 2 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 10 | 1 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 16 | 5 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 7 | 3 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 2 | 0 | 2
Hypoparathyroidism (Endocrine disorders) | 5 | 2 | 0 | 0
Blepharitis (Eye disorders) | 8 | 4 | 0 | 0
Cataract (Eye disorders) | 11 | 2 | 0 | 1
Corneal Toxicity (Eye disorders) | 0 | 2 | 0 | 0
Diplopia (Eye disorders) | 4 | 0 | 0 | 1
Dry Eye (Eye disorders) | 50 | 9 | 9 | 1
Eye Discharge (Eye disorders) | 0 | 2 | 0 | 0
Keratitis (Eye disorders) | 14 | 4 | 0 | 2
Lacrimation Increased (Eye disorders) | 11 | 3 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 6 | 1 | 1 | 1
Ulcerative Keratitis (Eye disorders) | 2 | 0 | 1 | 1
Vision Blurred (Eye disorders) | 28 | 5 | 3 | 0
Visual Acuity Reduced (Eye disorders) | 3 | 3 | 0 | 0
Xerophthalmia (Eye disorders) | 4 | 2 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 7 | 3 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 33 | 5 | 3 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 15 | 4 | 4 | 1
Angular Cheilitis (Gastrointestinal disorders) | 6 | 2 | 1 | 1
Ascites (Gastrointestinal disorders) | 8 | 3 | 2 | 0
Cheilitis (Gastrointestinal disorders) | 5 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 67 | 14 | 10 | 2
Diarrhoea (Gastrointestinal disorders) | 127 | 28 | 28 | 7
Dry Mouth (Gastrointestinal disorders) | 106 | 19 | 24 | 3
Dyspepsia (Gastrointestinal disorders) | 9 | 4 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 21 | 2 | 3 | 1
Glossitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Glossodynia (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Lip Dry (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Mouth Ulceration (Gastrointestinal disorders) | 10 | 4 | 4 | 0
Nausea (Gastrointestinal disorders) | 44 | 9 | 11 | 4
Stomatitis (Gastrointestinal disorders) | 122 | 26 | 22 | 3
Vomiting (Gastrointestinal disorders) | 40 | 7 | 11 | 3
Asthenia (General disorders) | 30 | 5 | 7 | 1
Fatigue (General disorders) | 63 | 10 | 16 | 1
Gait Disturbance (General disorders) | 4 | 1 | 1 | 1
Hyperthermia (General disorders) | 1 | 1 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 7 | 2 | 4 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0 | 1 | 1
Oedema Peripheral (General disorders) | 19 | 4 | 5 | 2
Pyrexia (General disorders) | 22 | 4 | 2 | 1
Hepatic Cytolysis (Hepatobiliary disorders) | 7 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 12 | 6 | 2 | 0
Conjunctivitis (Infections and infestations) | 15 | 5 | 3 | 0
Nail Bed Infection (Infections and infestations) | 0 | 0 | 1 | 2
Onychomycosis (Infections and infestations) | 5 | 1 | 1 | 1
Oral Candidiasis (Infections and infestations) | 6 | 1 | 3 | 1
Oral Herpes (Infections and infestations) | 5 | 0 | 0 | 1
Paronychia (Infections and infestations) | 43 | 7 | 5 | 2
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1
Skin Infection (Infections and infestations) | 4 | 3 | 0 | 1
Tinea Pedis (Infections and infestations) | 1 | 2 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 19 | 5 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 1 | 1 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 63 | 12 | 17 | 4
Aspartate Aminotransferase Increased (Investigations) | 59 | 12 | 12 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 34 | 3 | 4 | 1
Blood Chloride Decreased (Investigations) | 3 | 1 | 0 | 1
Blood Creatinine Increased (Investigations) | 21 | 3 | 2 | 0
Blood Phosphorus Increased (Investigations) | 20 | 1 | 2 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 11 | 2 | 0 | 1
Thyroxine Free Decreased (Investigations) | 1 | 0 | 0 | 1
Vitamin D Decreased (Investigations) | 1 | 0 | 0 | 1
Weight Decreased (Investigations) | 29 | 6 | 8 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 59 | 8 | 20 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 21 | 4 | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 3 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 156 | 29 | 42 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 | 2 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 4 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 3 | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 | 3 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 5 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 19 | 4 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 8 | 7 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 26 | 5 | 8 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 0 | 1 | 1
Fracture Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 10 | 3 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 7 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 5 | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 25 | 6 | 3 | 5
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Tendon Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Ageusia (Nervous system disorders) | 4 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 10 | 3 | 3 | 0
Dysgeusia (Nervous system disorders) | 37 | 11 | 5 | 0
Facial Paresis (Nervous system disorders) | 1 | 1 | 0 | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 24 | 3 | 4 | 3
Hypoaesthesia (Nervous system disorders) | 9 | 1 | 2 | 1
Neuralgia (Nervous system disorders) | 1 | 1 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 13 | 1 | 2 | 1
Seizure (Nervous system disorders) | 6 | 0 | 0 | 1
Taste Disorder (Nervous system disorders) | 8 | 1 | 5 | 0
Vith Nerve Disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 7 | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 14 | 2 | 5 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 6 | 2 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 4 | 1 | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 1 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39 | 10 | 4 | 3
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 16 | 4 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 15 | 1 | 2 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 44 | 13 | 6 | 2
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 77 | 12 | 9 | 1
Erythema (Skin and subcutaneous tissue disorders) | 7 | 3 | 2 | 0
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Hair Texture Abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Nail Discolouration (Skin and subcutaneous tissue disorders) | 32 | 4 | 9 | 3
Nail Disorder (Skin and subcutaneous tissue disorders) | 41 | 8 | 3 | 1
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 23 | 4 | 0 | 1
Nail Pigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Nail Ridging (Skin and subcutaneous tissue disorders) | 11 | 1 | 0 | 2
Nail Toxicity (Skin and subcutaneous tissue disorders) | 10 | 3 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 40 | 10 | 7 | 3
Onychomadesis (Skin and subcutaneous tissue disorders) | 18 | 3 | 3 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 73 | 17 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 3 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 18 | 8 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 1
Hypotension (Vascular disorders) | 13 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT04083976/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT04083976/SAP_001.pdf